CLINICAL TRIAL: NCT03310775
Title: The Effect of Korean Version of PEERS Social Skills Training for Young Adults (PEERS-YA-K) With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: B-1611-371-303
Record Dates: First submitted 2017-07-12; First posted 2017-10-16 (Actual); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2016-11

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Social skill training; PEERS
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case group (Experimental): Behavioral: parent-assisted social skills training program for young adults with autism spectrum disorder The subjects will participate in the treatment program weekly for a total of 14 weeks. The final visit will be made at the point three months after the completion of treatment to see mid- and long-term effects.
  Interventions: Behavioral: Parent-assisted social skills training program for young adult with ASD
- waitlist control group (Experimental): For this group, same intervention with the Experimental group will be provided after waiting for 16 weeks.
  Behavioral: Delayed intervention Intervention is provided to Waitlist Control Group after waiting for 16 weeks
  Interventions: Behavioral: Parent-assisted social skills training program for young adult with ASD

INTERVENTIONS:
Behavioral: Parent-assisted social skills training program for young adult with ASD — The subjects will participate in the treatment program weekly for a total of 16 weeks. The final visit will be made at the point four months after the completion of treatment to see long-term effects.
  Other Names: PEERS

SUMMARY:
Despite the psychosocial difficulties common among young adults with autism spectrum disorders(ASD), little to no evidence-based social skills interventions exist for this population. Using a randomized controlled trial(RCT) design, the current study tested the effectiveness of an evidence-based, caregiver-assisted social skills intervention known as PEERS for Young Adults with high-functioning young adults with ASD using self- and caregiver-report measures.

DETAILED DESCRIPTION:
1. Both the case and the control of this study shall be a high-functioning group consisting of young adults aged 18 to 35 years with ASD and an IQ of 70 or over. A total of 48 young adults will be recruited and divided into two groups. One will be the case group and the other will be the waitlist control group. And the study will be going on 3 institutions. Again, the case will be divided into two sub-groups of ten and carry out this new developed program for both parents and young adult. That is, the program will be carried out two times in each of both groups. The waitlist control group will be allowed to receive personal outpatient treatment and general therapeutic intervention from community while waiting.
2. Effects of the program will be measured both at the case and the control by using a scale which measures social interaction, quality of peer relationship, disposition of autism and social anxiety. Equal assessments for both the case and the control will be conducted right before the beginning of the program and right after the completion of the program and four months after the completion of the program.

ELIGIBILITY:
Inclusion Criteria:

* 18~35 years of age with ASD and IQ of 70 or over

Exclusion Criteria:

* Young adults who are hard to understand the content of treatment and carry out the task due to their IQs or limited linguistic abilities
* Young adults who are uncooperative in the treatment, lack motives and are hard to participate voluntarily
* Young adults who have behavior problems so clinically significant that they affects the therapeutic procedure or problems in controlling their emotion and have psychotic symptoms

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh M, Laugeson E, Kim JH, Lee K, Kim J, Lee S, Lim B, Cha S, Bong G, Yoon NH, Bahn GH, Yoo HJ. A Randomized Controlled Trial of the Korean Version of the Program for the Education and Enrichment of Relational Skills for Young Adults (PEERS(R)-YA-K) With Autism Spectrum Disorder: A Pilot Study. Front Psychiatry. 2021 Oct 6;12:730448. doi: 10.3389/fpsyt.2021.730448. eCollection 2021. PMID 34690837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited from the Child and Adolescent Psychiatric Clinic at Seoul National University Bundang Hospital, through advertisements at the Smile Together Foundation (a local advocacy institute of ASD), a community of child and adolescent psychiatrists, an internet group of families of youth with ASD.
Pre-assignment Details: Ten participants were excluded during the randomization procedure; six were not adequately motivated, one did not meet the diagnosis of ASD, one had difficulty understanding self-report scales, one had a problem with school, and one had to fulfill a military commitment.
Groups:
- Waitlist Control Group: For this group, same intervention with the Experimental group will be provided after waiting for 16 weeks.
  Behavioral: Delayed intervention Intervention is provided to Waitlist Control Group after waiting for 16 weeks
  Parent-assisted social skills training program for young adult with ASD: The subjects will participate in the treatment program weekly for a total of 16 weeks. The final visit will be made at the point four months after the completion of treatment to see long-term effects.
Period: Overall Study
Arm/Group | Case Group | Waitlist Control Group
Started | 19 | 18
Completed | 17 | 14
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — aggravation of depression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Case Group | Waitlist Control Group | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (3.7) | 23.5 (4.1) | 23.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 19 | 17 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 19 | 18 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Autism Diagnostic Observation Schedule(ADOS) at 4 Month
Description: The ADOS is a play-based, semistructured, standardized assessment of communication, social interaction, and play (i.e. imaginative use of materials) for individuals with a suspected diagnosis of autism or ASD. The ADOS consists of four modules, each of which can be selected on the basis of the participant's expressive language skills and hronological age. Module 4 of the ADOS is designed for adolescents and adults with fluent speech, and includes 10 essential and 5 optional activities. The scores from each activity are coded as well as those for five subdomains: language and communication, reciprocal social interaction, imagination, stereotyped behaviors and restricted interests, and other abnormal behaviors.
  minimum 0, maximum 18, higherscores mean a worse outcome.
Time Frame: baseline, after the completion of the treatment, 4 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Waitlist Control Group
Number analyzed (Participants) | 17 | 14
score on a scale
  communication | 3.3 (1.0) | 3.6 (1.3)
  social interaction | 7.5 (2.1) | 8.8 (2.3)
  Stereotyped behaviors and restricted interests | 1.0 (0.2) | 1.1 (0.2)
  Imagination | 0.4 (0.6) | 0.6 (0.1)

2. Primary Outcome: Change From Baseline in Test of Young Adult Social Skills Knowledge(TYASSK) at 4 Month
Description: The TYASSK is a 22-item criterion-referenced test developed for this study to assess the teen's knowledge about the specific social skills taught during the intervention. Two items were derived from key elements of each of the 11 didactic lessons. Teens were presented with sentence stems and asked to choose the best option from two possible answers. Scores range from 0 to 22, with higher scores reflecting greater knowledge of teen social skills.
Time Frame: baseline, 4 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Waitlist Control Group
Number analyzed (Participants) | 17 | 14
score on a scale | 17.5 (4.3) | 21.7 (3.4)

3. Primary Outcome: Change From Baseline in Korean Version of the Social Skills Rating System (K-SSRS) at 4 Month
Description: The SSRS consists of 38-items and took approximately 10 min to complete. Questionnaires were completed independently by the teen's parent and teacher. For example, items included ''Starts conversations rather than waiting for someone to talk first.'' The items were rated as either ''Never,'' ''Sometimes,'' or ''Very Often.'' The Social Skills and Problem Behaviors scales were derived from factor analysis.
  minimum 50 and maximum 163, and higherscores mean a better outcome
Time Frame: baseline,4 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Waitlist Control Group
Number analyzed (Participants) | 17 | 14
score on a scale | 115.7 (32.5) | 108.4 (26.3)

4. Primary Outcome: Change From Baseline in Social Responsiveness Scale-2 (SRS-2) at 4 Month
Description: The SRS is a 65-item questionnaire that assesses the various dimensions of interpersonal behavior, communication, and repetitive/stereotypic behavior that are characteristics of ASD.
  minimum 92, maximum 200, higherscores mean a worse outcome
Time Frame: baseline,4 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Waitlist Control Group
Number analyzed (Participants) | 17 | 14
score on a scale | 146.5 (22.9) | 147.9 (24.3)

5. Secondary Outcome: Korean Version of the Vineland Adaptive Behavior Scale, Second Edition
Description: The K-VABS is an interviewed survey and measures adaptive behaviors of individuals such as personal and social skills, used for everyday living from birth to age 90. These are based on the reports of primary caregivers and teachers. The K-VABS contains 5 domains each with 2-3 subdomains. The main domains are: Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior (optional). Behaviors are rated on a 0 (a skill that is not used by the individual) - 2 (a skill used most of the time) rating scale. The current study used only the communication, daily living skills, and socialization domains.
  minimum 25, maximum 108, higherscores mean a better outcome.
Time Frame: baseline,4 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Waitlist Control Group
Number analyzed (Participants) | 17 | 14
score on a scale
  communication | 75.0 (13.4) | 70.5 (16.4)
  daily living skills | 78.3 (16.5) | 74.4 (20.9)
  socialization | 71.9 (18.3) | 65.9 (12.7)

6. Secondary Outcome: Change From Baseline in Beck Depression Inventory (BDI) at 4month
Description: The BDI consists of 21 items measuring the severity of subjective symptoms of depression, with emotional, cognitive, motivational, and physiological symptom profiles for adults. Each question has four possible answer choices, scored from 0 (no symptoms) to 3 (the most severe symptoms).
  minimum 1, maximum 45, higherscores mean a worse outcome
Time Frame: baseline,4 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Case Group | Waitlist Control Group
Number analyzed (Participants) | 17 | 14
score on a scale | 12.8 (10.2) | 14.5 (11.4)

ADVERSE EVENTS:
Time Frame: no adverse event through study completion, an average of 1 year
Arm/Group | Case Group | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT03310775/Prot_SAP_000.pdf